CLINICAL TRIAL: NCT00833196
Title: An International, Observational Study to Define Factors Influencing Response to One BoNT-A Injection Cycle in Subjects Suffering From Idiopathic Cervical Dystonia
Brief Title: Factors Influencing Response to One BoNT-A Injection Cycle in Subjects Suffering From Idiopathic Cervical Dystonia
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: Y-79-52120-131
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Idiopathic Cervical Dystonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A post marketing, international, multicenter, observational, prospective, longitudinal study. The purpose of the study is to describe cervical dystonia sub-types with their injection protocols and response to BoNT-A.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic cervical dystonia
* TWSTRS severity score ≥ 15
* At least a 12-week interval between the last injection (BoNT-A or BoNTB) and inclusion
* Written informed consent prior to collect the data

Exclusion Criteria:

* Contraindications to any BoNT-A preparations
* Secondary cervical dystonia
* Subject already been included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic cervical dystonia
Sampling Method: Non-Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Responder rate at peak effect following one BoNT-A injection cycle without any deviations from routine practice | Around 4 weeks post injection

SECONDARY OUTCOMES:
To describe TWSTRS change scores from inclusion (total score & subscales scores) | Baseline, and around 4 weeks and 3 months post injection
To describe tremor change score from inclusion (TSUI scale) | Baseline, and around 4 weeks and 3 months post injection
To describe the Cervical Dystonia Impact Profile (CDIP) 58 change from inclusion | Baseline, and around 4 weeks post injection
To describe subject and investigator's CGI scores | Around 4 weeks post injection
To identify prognostic factors for response (Exploratory Objective) | baseline, and around 4 weeks and 3 months post injection

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (39):
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown
  - St Vincent's Hospital, Fitzroy
  - Austin Hospital, Heidelberg
  - Westmead Hospital, Penrith
  - Alfred Hospital, Prahran
- Belgium (5):
  - AZ Sint Jan Brugge, Bruges
  - UZ Gent, Ghent
  - Leuven
  - Centre Hospitalier de Liège, Domaine Universitaire Sart Tilmen, Liège
  - AZ Sint Augustinus Wilrijk, Wilrijk
- Czechia (4):
  - Fakultní nemocnice U Sv.Anny, Brno
  - Fakultní nemocnice Olomouc, Olomouc
  - Krajská nemocnice Pardubice, Pardubice
  - Všeobecná fakultní nemocnice, Prague
- France (7):
  - Hôpital Neurologique et Neurochirurgical Pierre Wertheimer, Bron
  - Hôpital Roger Salengro, Lille
  - Hôpital La Timone, Marseille
  - Hôpital Pasteur - CHU Nice, Nice
  - Hôpital La Pitié Salpétrière, Paris
  - Hôpital Haut Lévêque, Pessac
  - Hôpital Purpan, Toulouse
- Germany (6):
  - Praxis für Neurologie, Berlin
  - Praxis für Neurologie, Bochum
  - Praxis für Neurologie, International Neuroscience Institute, Hanover
  - Praxis für Neurologie, Neusaß
  - Praxis für Neurologie und Psychatrie, Schorndorf
  - Krankenhaus der Barmherzigen Brüder, Trier
- Netherlands (2):
  - Martini Ziekenhuis Groningen, Groningen
  - Tergooiziekenhuizen Hilversum, Hilversum
- Portugal (3):
  - Hospital Santa Maria, Lisbon
  - Hospital General San Antonio - Centro Hospitalar do Porto, Porto
  - Serviço de Neurologia - Hospital de São João, Porto
- Russia (4):
  - 16, ulitsa Vorovskogo, Chelyabinsk
  - 12a, ulitsa Karbyisheva, Kazan'
  - 80, Volokolamskoye shossee, Moscow
  - 6/8, ulitsa L'va Tolstogo, Saint Petersburg
- United Kingdom (3):
  - Royal Devon & Exeter Hospital, Exeter
  - National Hospital for Neurology & Neurosurgery, London
  - Walton Centre for Neurology & Neurosurgery, Hope Hospital, Manchester

REFERENCES:
- [Derived] Trosch RM, Misra VP, Maisonobe P, Om S. Impact of abobotulinumtoxinA on the clinical features of cervical dystonia in routine practice. Clin Park Relat Disord. 2020 Jun 15;3:100063. doi: 10.1016/j.prdoa.2020.100063. eCollection 2020. PMID 34316644
- [Derived] Misra VP, Ehler E, Zakine B, Maisonobe P, Simonetta-Moreau M; INTEREST IN CD group. Factors influencing response to Botulinum toxin type A in patients with idiopathic cervical dystonia: results from an international observational study. BMJ Open. 2012 Jun 14;2(3):e000881. doi: 10.1136/bmjopen-2012-000881. Print 2012. PMID 22700836